CLINICAL TRIAL: NCT02071485
Title: Non-Invasive Brain-Computer Interface for Virtual Object Control
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1312M46726
Record Dates: First submitted 2014-02-18; First posted 2014-02-26 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Individuality

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: Subjects in this study will receive no treatment and rather will only be trained in using the motor imagination-based BCI system

SUMMARY:
A brain-computer interface (BCI) is a system that provides a separate output pathway for neurological signals whereby they can be interpreted to determine the user's intended cognitive action. Utilizing EEG-based sensorimotor rhythms (SMRs) generated in the motor cortex has allowed subjects to control virtual computer cursors in up to three dimensions by simply imagining the movement of a specified body part. Nevertheless, the scalp EEG signals are smeared by the volume conduction effect and measurement noise. The overall hypothesis of this study is that EEG-based virtual object control may help reveal optimal motor imagination tasks best used in a BCI.

The PI's hypotheses include: (1) The use of advanced signal processing techniques will better reveal characteristics of EEG signals that represent the underlying motor cognitive function of the subject; (2) BCI systems based on SMR generated using motor imaginations will allow effective control of a virtual object in real time; (3) EEG imaging techniques will provide insight into the areas of cortical activation during a motor imagery task that can be utilized to increase the spatial resolution of non-invasive BCI's.

DETAILED DESCRIPTION:
The goal of the present study is to explore advanced signal processing techniques that will better reveal characteristics of EEG signals that represent the underlying motor cognitive function of the subject, and conduct experiments to better control an virtual object on the computer screen including a cursor or a helicopter.

The primary objective of this study is to test the above hypotheses (1) and (2) in a healthy subject population.This study will determine the ability of subjects with full cognitive function to control a non-invasive brain-computer interface by imagining a particular movement. Using non-invasive methods, we will investigate the neural processes that occur during the motor imagination tasks associated with controlling a virtual object. Using a variety of motor imaginations, we will determine which tasks are best used for BCI control by quantitative means of BCI performance and neurological dynamic system analysis.

Subjects for this study will be healthy, English speaking adult volunteers (18-64 years old) with no history of mental illness, neurological deficit, or traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Between the age of 18 and 64

Exclusion Criteria:

* History of traumatic brain injury/brain lesion, neurological deficit or neurodegenerative disorder

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Students and workers at the University of Minnesota - Twin Cities campus
Sampling Method: Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2014-03; Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
Classification accuracy (%) and Cohen's Kappa Coefficient (unit-less) will be measured by discriminating features within the EEG time courses of different motor imagery tasks. | two years

CONTACTS AND LOCATIONS:
Overall Officials: Bin He, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Nils Hasselmo Hall at the University of Minnesota - Twin Cities campus, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided